CLINICAL TRIAL: NCT06372977
Title: Kappa Index Versus Csf Oligoclonal Bands in Diagnosis of Multiple Sclerosis and Prediction of Disease
Brief Title: Kappa Index Versus Csf Oligoclonal Bands in Diagnosis of ms and Prediction of Disease Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham mohamed ahmed abdelsater, doctor, Assiut University
Other Study IDs: kappa index in ms
Record Dates: First submitted 2024-03-30; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: (-ve OCB )(70 patients) Control group which include patients with inflammatory and non-inflammatory neurological diseases (such as cerebral small vessel disease or unspecific white matter lesion )
  Interventions: Diagnostic Test: kappa index
- 2: (+ve OCBs )(70 patients) Patients presenting for the diagnostic workup, including CSF analysis , of clinical and/or MRI suspicion of MS or CIS.
  Interventions: Diagnostic Test: kappa index

INTERVENTIONS:
Diagnostic Test: kappa index — CSF albumin /serum albumin ratio (Qalb) k-index = (CSF kFLC/serum kFLC)/Qalb

SUMMARY:
To:

1. Compare the diagnostic performance of cerebrospinal fluid kappa index to that of cerebrospinal fluid IgG oligoclonal bands in differentiating multiple sclerosis from other inflammatory and non-inflammatory neurological diseases .
2. Assess the role of kappa free light chain and oligoclonal bands in predicting disease activity (conversion from clinical isolated syndrome to multiple sclerosis)

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic inflammatory immune-mediated disorder of the central nervous system.Diagnosis requires the combination of clinical signs and symptoms with paraclinical findings obtained by magnetic resonance imaging and cerebrospinal fluid analysis .which are componants of the 2017 McDonald criteria .So far, the gold standard for demonstrating intrathecal IgG synthesis is represented by selective oligoclonal bands in cerebrospinal fluid by isoelectric focusing (IEF), alongside an elevated IgG index .However, the detection of oligoclonal bands in cerebrospinal fluid has several limits as , it requires a time-consuming and expensive laboratory technique, with about three hours needed to obtain results Furthermore, it only provides aqualitative information about the presence of IgG in CSF .During CNS inflammation , kappa free light chain are secreted in the CSF and their concentration reflect the degree of intrathecal B cells and plasma cells activation .Measurement of KFLC could help diagnosis of OCB negative MS and identify intrathecal immunoglobulin synthesis in patient presenting with one isolated band on isoelectric focusing , and it is fully automated,rater independent, stable against preanalytical errors . Thus, the intrathecal synthesis of free light chains are more sensitive, less costly, and less time-consuming compared To OCB detection .The most reliable parameter used to assess FLC diagnostic value in MS is the k-index, .So κ-FLC index predicted the time to conversion to MS as well as disability progression . So patients with early MS and high κ-FLC index is an independent risk factor for conversion from CIS to MS

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CIS or MS according to the 2017 revision of the McDonald criteria
* Patients diagnosed with RIS (Radiological isolated syndrome) according to the criteria by Okuda
* Age between 18 and 40 years.

Exclusion Criteria:

* History of exposure, in the 30 days prior to CSF collection, to immunosuppressant or immunomodulatory therapies .
* Peripheral neurological disorders .
* Infectious CNS disease.
* CNS tumor.
* Monoclonal gammopathy .
* Chronic kidney injury (GFR <30 ml /min/1.75m2 )

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: we will select for this study 140 patients including control group and patients group aged between 18 -40
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assess the diagnostic performance of CSF k index in differentiating MS from other inflammatory and non-inflammatory neurological diseases . | baseline
  measure specificity and sensitivity of kappa free light chain
Assess the diagnostic performance of CSF IgG OCBs in differentiating MS from other inflammatory and non-inflammatory neurological diseases . | baseline
  measure specificity and sensitivity of cerebrospinal fluid oligoclonal bands

SECONDARY OUTCOMES:
Assess the role of k FLC in predicting disease activity (conversion from CIS to MS) | baseline
  measure positive predictive value and negative predictive value of kappa free light chain
Assess the role of OCBs in predicting disease activity (conversion from CIS to MS) | baseline
  measure positive predictive value and negative predictive value of oligoclonal bands

REFERENCES:
- [Background] Gaetani L, Di Carlo M, Brachelente G, Valletta F, Eusebi P, Mancini A, Gentili L, Borrelli A, Calabresi P, Sarchielli P, Ferri C, Villa A, Di Filippo M. Cerebrospinal fluid free light chains compared to oligoclonal bands as biomarkers in multiple sclerosis. J Neuroimmunol. 2020 Feb 15;339:577108. doi: 10.1016/j.jneuroim.2019.577108. Epub 2019 Nov 7. PMID 31743879
- [Background] Duell F, Evertsson B, Al Nimer F, Sandin A, Olsson D, Olsson T, Khademi M, Hietala MA, Piehl F, Hansson M. Diagnostic accuracy of intrathecal kappa free light chains compared with OCBs in MS. Neurol Neuroimmunol Neuroinflamm. 2020 Jun 11;7(4):e775. doi: 10.1212/NXI.0000000000000775. Print 2020 Jul. PMID 32527760